CLINICAL TRIAL: NCT05665192
Title: Real-World Clinical and Patient Reported Outcomes With Fedratinib for Myelofibrosis Post-Ruxolitinib
Brief Title: A Study to Assess Real-World Patient-Reported Outcomes With Fedratinib for Myelofibrosis Post-Ruxolitinib
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA054-1014
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Myelofibrosis
Keywords: Primary Myelofibrosis; Thrombocythemia Myelofibrosis; Fedratinib; Ruxolitinib
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1: Participants that have discontinued RUX therapy and initiated FEDR prospectively

SUMMARY:
The purpose of this study is to determine real-world patient-reported outcomes with fedratinib (FEDR) therapy for myelofibrosis (MF) in the real-world (RW) setting.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Primary myelofibrosis (PMF), post- Essential thrombocythemia (ET) Myelofibrosis (MF), or post- Polycythemia vera (PV) MF
* Treated with FEDR and initiated treatment after 16 August 2019.
* Received prior treatment with RUX.
* Had spleen assessed at time of initiation of FEDR by palpation.
* Able to read and speak English
* Willing to provide informed consent
* Willing to provide permission to the site to release her/his medical information to the study investigators according to the study-specific eCRF
* Willing to complete the baseline survey prior to first FEDR

Exclusion Criteria:

* Past or current participant in any FEDR-related clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of participants who have discontinued RUX and will be initiating FEDR prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Percentage change in Total Symptom Score (TSS) assessed by Myelofibrosis Symptom Assessment Form (MFSAF) | Percentage change in Total Symptom Score (TSS) assessed by Myelofibrosis Symptom Assessment Form (MFSAF)
Absolute change in TSS assessed by MFSAF | At Baseline, 3 and 6 months post-FEDR initiation
Proportion of participants reporting individual symptoms in TSS assessed by MFSAF | At Baseline, 3 and 6 months post-FEDR initiation
Severity of each reported symptom in TSS assessed by MFSAF | At Baseline, 3 and 6 months post-FEDR initiation
Frequency of report of domain assessed by Patients' Global Impression of Change (PGIC) | At Baseline, 3 and 6 months post-FEDR initiation
Absolute reduction assessed by Patient-Reported Outcomes Measurement Information System Global-10 (PROMIS-10) | At Baseline, 3 and 6 months post-FEDR initiation

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Cardinal Health Specialty Solutions, Dublin, Ohio, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html